CLINICAL TRIAL: NCT05983276
Title: Combination of the Hypomethylating Agent Decitabine and the Nuclear Export Receptor XPO-1 Inhibitor Selinexor to Reverse Platinum Resistance in Relapsed/Refractory Epithelial Ovarian Cancer
Brief Title: Decitabine and Selinexor in Combination to Reverse Drug Resistance With Standard Chemotherapy in Ovarian Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Loyola University (Other)
Collaborators: Karyopharm Therapeutics Inc (Industry)
Responsible Party: Principal Investigator, Patrick Stiff, Senior Professor, Loyola University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 215615
Record Dates: First submitted 2023-07-12; First posted 2023-08-09 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Ovarian Cancer
Keywords: Ovarian Cancer; Platinum Resistance; Relapsed/Refractory Epithelial; Fallopian Tube; Primary Peritoneal Cancer
MeSH Terms: conditions — Ovarian Neoplasms; Recurrence | interventions — Decitabine; Carboplatin; Paclitaxel; Albumin-Bound Paclitaxel; selinexor

STUDY DESIGN:
Intervention Model Description: Once selected for therapy, the participant will receive the following treatment in the outpatient setting:
  Days 1-5: Decitabine 10 mg; m2 IV daily Day 6: carboplatin AUC 5 and paclitaxel 80 mg; m2 Days 13, 20, and 27: paclitaxel 80 mg/m2 For a single 28 day cycle.
  Assess Response toxicities and immune effector cell changes.
  Days 1-5: Decitabine 10 mg/m2 IV daily; Day 6: carboplatin AUC 5 and paclitaxel 80 mg/ m2; Day 7 and weekly thereafter (day 14, 21, 28, 35…) Selinexor 60 mg PO Days 13, 20, and 27: paclitaxel 80 mg/m2 each given x five 28 day cycles
  Assess responses by exam, CT scan and blood tests, assess toxicities, and immune effector cell changes as well as progression and overall survival
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Decitabine / Selinexor/ Carboplatin / Paclitaxel (Experimental): C1:
  Days 1-5: Decitabine 10 mg/m2 IV daily Day 6: carboplatin AUC 5 and paclitaxel 80 mg/ m2 Days 13, 20, and 27: paclitaxel 80 mg/m2 For a single 28 day cycle
  Assess Response toxicities and immune effector cell changes
  C2-C6:
  Days 1-5: Decitabine 10 mg/m2 IV daily Day 6: carboplatin AUC 5 and paclitaxel 80 mg/ m2 Day 7 and weekly thereafter (day 14, 21, 28, 35…) Selinexor 60 mg PO Days 13, 20, and 27: paclitaxel 80 mg/m2 each given x five 28 day cycles
  Assess responses by exam, CT scan and blood tests, assess toxicities, and immune effector cell changes as well as progression and overall survival
  Interventions: Drug: Decitabine; Drug: Carboplatin; Drug: Paclitaxel; Drug: Selinexor

INTERVENTIONS:
Drug: Decitabine — Decitabine is classified as hypomethylation agents. It works by helping the bone marrow produce normal blood cells and by killing abnormal cells in the bone marrow.
  Other Names: Dacogen
Drug: Carboplatin — Carboplatin is classified as an alkylating agent that is used to treat ovarian cancer.
  Other Names: Paraplatin
Drug: Paclitaxel — Paclitaxel is classified as a "plant alkaloid," a "taxane" and an "antimicrotubule agent."
  Other Names: Abraxane
Drug: Selinexor — Selinexor is in a class of medications called selective inhibitors of nuclear export (SINE). It works by killing cancer cells.
  Other Names: Xpovio, Nexpovio

SUMMARY:
The goal of this clinical trial is to learn about the side effects and effectiveness of this novel four-drug combination of chemotherapy (decitabine, selinexor, carboplatin and paclitaxel) on patients with relapsed ovarian, fallopian or primary peritoneal carcinoma.

Recently the investigators have found that the combination of decitabine and selinexor, two Food and Drug Administration (FDA) approved chemotherapy agents, may prevent or reverse the development of drug resistance and further the remissions and duration of remissions with standard ovarian cancer chemotherapy with carboplatin and paclitaxel. As decitabine and selinexor are not FDA approved for the participant's cancer, these agents are investigational.

DETAILED DESCRIPTION:
Participants enrolled in this study protocol will receive therapy with decitabine followed by usual doses of carboplatin and paclitaxel for one cycle. If the participant tolerates this well, the selinexor will be added to the second and subsequent cycles of therapy given at 4-week intervals, in the out-patient setting. The participant will be asked to complete 9 study visits during their active therapy during each cycle: Days 1-5 of each cycle the participant will receive decitabine treatments over 1 hour, with carboplatin and paclitaxel given on day 6. Paclitaxel alone will continue weekly for 3 weeks on days 13, 20 and 27 of the 28-day cycle. The 5 days of daily decitabine therapy lasts about 1 hour and the carboplatin and paclitaxel treatment last 4 hours, with single agent paclitaxel being only 1 hour.

Selinexor is not added until cycle 2 and is given orally weekly on days 7, 14, 21, and 28 of the 28-day cycle. Weekly clinic visits are required for the first two cycles at the time paclitaxel is administered.

The participant's progress will be assessed and if a remission is achieved the participant would continue the therapy for up to 6 cycles.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be greater than or equal to 18 years of age
* Participants must have an Eastern Cooperative Oncology Group (ECOG) Performance Status PS less than or equal to 2.
* Participants must have histological or cytological proven epithelial ovarian cancer, fallopian tube or primary peritoneal carcinoma with relapse or disease progression after prior treatment by exam, computed tomography (CT), PET/CT, or magnetic resonance imaging (MRI) may be enrolled. All cell types including clear cell carcinoma are eligible.
* Participants must have failed or relapsed after a platinum and taxane containing combination
* Participants must have adequate hepatic function
* Participants must have adequate renal function
* Participants must be able to swallow and retain oral medications
* Participants must have measurable disease according to Gynecologic Cancer Intergroup CA125 criteria
* Participants with stable (for 2 months or longer), treated (by radiotherapy) CNS metastases are eligible
* Participants with active hepatitis B virus (Hep B) are allowed if antiviral therapy for hepatitis B has been given for greater than 8 weeks.

Exclusion Criteria:

* Participants must not have received Selinexor or another XPO1 inhibitor previously.
* Participants must not have had any concurrent medical condition or disease (eg, uncontrolled active hypertension, uncontrolled active diabetes, active systemic infection, etc.)
* Participants must not have uncontrolled active infection. Participants on prophylactic antibiotics or with a controlled infection within 1 week prior to C1D1 are acceptable.
* Participants must not have known intolerance, hypersensitivity, or contraindication to platinum or taxane therapy
* Participants must not have active, unstable cardiovascular function
* Participants must not have myocardial infarction within 3 months prior to starting
* Participants with untreated central nervous system (CNS) metastases are ineligible.
* Participants must not have had prior chemotherapy or radiation therapy
* Participants must not have DVT related to metastatic disease requiring ongoing anticoagulation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-11-16 (Actual); Primary Completion 2030-08-28 (Estimated); Study Completion 2031-08-28 (Estimated)

PRIMARY OUTCOMES:
40 participants evaluated for safety with treatment-related adverse events and grading using CTCAE 4.3. | 6 months
  To determine the safety of two agents in combination to reverse platinum resistance in ovarian cancer: the hypomethylating agent, decitabine, and the nuclear export receptor XPO1 inhibitor, selinexor, combined with carboplatin and paclitaxel in patients with relapsed/refractory epithelial ovarian carcinoma

SECONDARY OUTCOMES:
40 participants evaluated to determine the clinical efficacy of this novel regimen in both platinum sensitive and resistant recurrent disease as measured by response rates. Response rates (partial response [PR] and complete response [CR]) | 6 months
  To determine the clinical efficacy of this novel regimen in both platinum sensitive and resistant disease as measured by response rates
40 participants evaluated to determine the cellular immune effects of this combination. B and T cell numbers and subsets after therapy. | 6 months
  This is an exploratory endpoint to determine if there is a potential immune enhancement of this combination on numbers of Immune T and B cells after therapy (15% or higher increase in cell numbers/mm3) when compared to pre-treatment values and whether this correlates to response rates.
40 participants evaluated for tolerability with treatment-related adverse events and grading using CTCAE 4.3. | 6 months
  To determine the tolerability of two agents that reverse platinum sensitivity in ovarian cancer, the hypomethylating agent, decitabine, and the nuclear export receptor XPO1 inhibitor, Selinexor, combined with carboplatin and Taxol in patients with relapsed/refractory epithelial ovarian carcinoma

CONTACTS AND LOCATIONS:
Overall Officials: Patrick L Stiff, MD, Principal Investigator — Loyola University
Locations (1):
- Loyola University Medical Center, Maywood, Illinois, United States